CLINICAL TRIAL: NCT05441293
Title: b Division of Plastic Surgery, Department of Surgery, Wan Fang Hospital, Taipei Medical University, Taipei, Taiwan
Brief Title: Determinants of the Success of Flap Reconstruction: Outcome Analysis of 484 Surgeries for Pressure Injury
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WanFangW2
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- debridements group: During study peroid, the patient who received debridement surgery for pressure injury
  Interventions: Procedure: flap reconstruction
- flap reconstructions group: During study peroid, the patient who received flap reconstruction surgery for pressure injury
  Interventions: Procedure: flap reconstruction

INTERVENTIONS:
Procedure: flap reconstruction — received flap reconstruction over sacrum, back, trochanter, ischium, elbow, and lower extremities

SUMMARY:
Background: Pressure injury (PI) mainly occurs in bedridden older adults or those with physical limitations. PI treatment is typically long-term, requiring coordination between health-care workers and the patient's caregiver. Here, we aimed to determine the appropriate timing to conduct flap reconstruction in patients with PIs and identify factors affecting surgical outcomes.

Materials and Methods: We retrospectively reviewed the data of all patients who received debridement or flap reconstruction surgery for PIs in our hospital from January 2016 to December 2021. The extracted data included patient demographics, surgical records, blood test results, vital signs, and flap outcomes. Next, these characteristics including the flap outcomes of our patients with PIs were analyzed, along with the risk factors for poor wound healing and complications.

ELIGIBILITY:
Inclusion Criteria:

all patients who received debridement or flap reconstruction surgery for Pressure injury in Wan Fang Hospital from January 2016 to December 2021

Exclusion Criteria:

the patients who did not received debridement or flap reconstruction surgery for Pressure injury

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who received debridement or flap reconstruction surgery for Pressure injury in Wan Fang Hospital from January 2016 to December 2021
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Complete wound healing | from January 2016 to December 2021
  no presentation of wound drainage or wound dehiscence at the surgical site 14 days after drainage tube removal.

IPD SHARING:
Plan to Share IPD: No
the data are not available for sharing.